CLINICAL TRIAL: NCT02887404
Title: Evaluation of Spine Surgery Analgesic Pathway: A Randomized Controlled Trial
Brief Title: Evaluation of Spine Surgery Analgesic Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kamal Maheshwari, MD MPH, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-012
Record Dates: First submitted 2016-08-17; First posted 2016-09-02 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Posterior Spine Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spine surgery analgesic pathway (Experimental): Before surgery the subject will be given one time oral dose Acetaminophen (1000 mg ) and gabapentin (600 mg).
  During surgery the subject will receive an infusion of ketamine (5 mcg/kg/min) and lidocaine (1.5 mg/kg/hr start before the incision and decreased to 1 mg/kg/hr at start of closing and continued to PACU and stop at the first oral intake).
  After surgery, the surgical team will manage pain medication and will consult acute pain management team as needed.
  Interventions: Other: Spine surgery analgesic pathway
- Usual care (Active Comparator): Placebo- Before surgery the subject will be given one time placebo oral dose Acetaminophen (1000 mg ) and gabapentin (600 mg).
  Placebo- During surgery the subject will receive a placebo infusion of - ketamine (5 mcg/kg/min) and lidocaine (1.5 mg/kg/hr start at incision and decreased to 1 mg/kg/hr at start of closing and continued to PACU and stop at the first oral intake).
  After surgery, the surgical team will manage pain medication and will consult acute pain management team as needed.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Spine surgery analgesic pathway — Enhanced pain management care
  Arms: Spine surgery analgesic pathway
Other: Usual Care — Standard of pain management care
  Arms: Usual care

SUMMARY:
Investigators plan to study the role of spine surgery analgesic pathways - for procedures with high risk of postoperative pain - in improving the quality of recovery

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing "spine surgery analgesic pathway" with "usual care" in improving postoperative quality of recovery and pain management in spine surgery patients. At the time of surgery office visit or at the time of preoperative assessment by anesthesia care team, risk factor for suboptimal pain management will be identified and documented. Patients will be assessed at the time for surgical office visit for their risk for severe post-operative pain. Patients with 2 or more risk factors will be classified as high-risk for severe postoperative pain and the patients with less than 2 factors as low risk. After obtaining informed consent spine surgery patients will be randomized 1:1 in one of the 2 study groups on the day of the surgery:

1. "Usual care" group A
2. "Care pathway" group B

If the participant is randomized to the "spine surgery analgesic pathway" group the participant will be evaluated by the Acute Pain Management Service (APMS) before the surgery for their specific pain management needs. The participant will also get some additional medication for pain in preoperative and intraoperative period. Before surgery the participant will receive Acetaminophen and Gabapentin pills. During the surgery, once the participant is asleep the participant will receive an infusion of ketamine and lidocaine through the participant venous line. After the surgery the participant will receive pain medications as per current standard protocol including acetaminophen and gabapentin. Pain management team specialist will follow for pain control after a surgery as needed.

If the participant is randomized to the "usual care" group the participant will be given placebo preoperatively; the rest of the time pain medication will be provided in a routine manner as per the anesthesia care team and the surgical team. Pain management team specialist will follow for pain control after a surgery as needed.

The primary outcome will be assessed on post-operative day 3: The participants will complete a short survey about quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old at time of surgery - Adult patients differ from pediatric patients in that adult spines are stiffer than pediatric patients.
* Posterior spine surgery
* Surgery performed at Cleveland Clinic main campus

Exclusion Criteria:

* Allergy or hypersensitivity to lidocaine, ketamine, acetaminophen, gabapentin
* Current or recent drug abuse (within past 6 months)
* Pregnancy
* Immune system disease such as HIV, AIDS
* Undergoing immunosuppressive treatment
* Recent history of sepsis
* Contraindications to lidocaine such as heart block and hepatic insufficiency
* Heart failure with ejection fraction less than 30%
* Liver dysfunction manifested with increased liver enzymes to double the normal and INR of 2 or higher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2016-07; Primary Completion 2019-01 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Study Chair — Department Chair
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Spine Surgery Analgesic Pathway: Before surgery, the subject will be given one-time oral dose Acetaminophen (1000 mg ) and gabapentin (600 mg).
  During surgery, the subject will receive an infusion of ketamine (5 ug/kg/min; Ketamine was stopped at wound closure.) and lidocaine (1.5 mg/kg/hr start before the incision and decreased to 1 mg/kg/hr at start of closing and continued to PACU and stop at the first oral intake).
  After surgery, the surgical team will manage pain medication and will consult acute pain management team as needed.
  Spine surgery analgesic pathway: Enhanced pain management care
- Usual Care: Placebo- Before surgery the subject will be given one time placebo oral dose Acetaminophen (1000 mg ) and gabapentin (600 mg).
  Placebo- During surgery the subject will receive a placebo infusion of - ketamine (5 mcg/kg/min) and lidocaine (1.5 mg/kg/hr start at incision and decreased to 1 mg/kg/hr at start of closing and continued to PACU and stop at the first oral intake).
  After surgery, the surgical team will manage pain medication and will consult acute pain management team as needed.
  Usual Care: Standard of pain management care
Period: Overall Study
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Started | 150 | 149
Completed | 150 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care | Total
Number analyzed (Participants) | 150 | 149 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12) | 63 (11) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 78 | 147
  Male | 81 | 71 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 144 | 140 | 284
  Black or African American | 5 | 6 | 11
  Other | 0 | 2 | 2
  Unknown | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (7) | 32 (7) | 31 (7)
Smoking [Count of Participants; unit: Participants] | 71 | 73 | 144
History of diabetes [Count of Participants; unit: Participants] | 33 | 25 | 58
History of chronic pain [Count of Participants; unit: Participants] | 120 | 108 | 228
Previous opioid use [Count of Participants; unit: Participants] | 80 | 81 | 161
High anxiety before surgery [Count of Participants; unit: Participants] | 54 | 54 | 108
Preoperative pain score [Mean (Standard Deviation); unit: units on a scale] — The preoperative pain score rages from 0-10 where 0 means no pain and 10 means the worst pain.
  units on a scale | 5.3 (2.8) | 5.3 (2.7) | 5.3 (2.8)
ASA status, No (%) [Count of Participants; unit: Participants] — ASA: American Society of Anesthesiologists Classification (ASA Class), which assesses a patient's overall health.
  I refer to ASA1-2 and II refer to ASA3 and III refer to ASA4-5.
  ASA1: Patient is a completely healthy fit patient.
  ASA2: Patient has mild systemic disease.
  ASA3: Patient has severe systemic disease that is not incapacitating.
  ASA4: Patient has incapacitating disease that is a constant threat to life.
  ASA5: A moribund patient who is not expected to live 24 hour with or without surgery.
  Participants
    I | 1 | 2 | 3
    II | 32 | 21 | 53
    III | 117 | 126 | 243
Charlson comorbidity index, No(%) [Count of Participants; unit: Participants] — The Charlson comorbidity index is a risk score assigned to patients for assessing their one-year mortality risk. It is based on a weighted count of specific chronic conditions in a patient's diagnosis history. Higher scores mean higher risk. Generally 0-2 means low risk; 3-4 means moderate risk and above 5 means high risk.
  Participants
    0 | 80 | 83 | 163
    1 | 36 | 34 | 70
    2 | 21 | 20 | 41
    3 | 4 | 7 | 11
    4 and above | 9 | 5 | 14
No. of risk factors for uncontrolled postoperative pain [Count of Participants; unit: Participants] — The risk factors for uncontrolled postoperative pain were defined in the protocol and included young age (60 yr old and younger), female sex, chronic pain for more than 3 months, high preoperative pain score (VAS scale ≥7), preoperative high anxiety level, and multilevel surgery.
  Participants
    1 | 3 | 0 | 3
    2 | 40 | 40 | 80
    3 | 44 | 42 | 86
    4 | 32 | 47 | 79
    5 | 26 | 18 | 44
    6 | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery
Description: Assessment of postoperative recovery should be multidimensional including physiological parameters, functional recovery parameters, and patient-reported outcomes. Quality of postoperative recovery will be assessed by asking the patient "how have you been feeling during the past 24 hours." Using the Quality of recovery form (QoR15) to document their replies. Quality of recovery (QoR15) score of (0 to 10), where: (0) none of the time (poor) and (10) equal all of the time (excellent). There are a total of 15 questions with each score ranging from 0 to 10. The range of reported total score is 0-150 where higher scores mean better quality of recovery.
Time Frame: Three days after surgery
Population: 21 patients in the treatment group were missing and 20 patients were missing in the placebo group
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Spine Surgery Analgesic Pathway: Before surgery the subject will be given one time oral dose Acetaminophen (1000 mg ) and gabapentin (600 mg).
  During surgery the subject will receive an infusion of ketamine (5 mcg/kg/min) and lidocaine (1.5 mg/kg/hr start before the incision and decreased to 1 mg/kg/hr at start of closing and continued to PACU and stop at the first oral intake).
  After surgery, the surgical team will manage pain medication and will consult acute pain management team as needed.
  Spine surgery analgesic pathway: Enhanced pain management care
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 129 | 129
units on a scale | 109 (25) | 109 (23)
Statistical Analysis 1: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Superiority; p = 0.92, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-6 to 6]

2. Secondary Outcome: Opioid Utilization
Description: Opioid consumption within the initial 48 h was converted to IV morphine equivalents using the conversions specified in Supplemental Digital Content 1 (http:// links.lww.com/ALN/C178).
Time Frame: up to 48 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
mg | 72 [48 to 113] | 75 [50 to 152]
Statistical Analysis 1: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Non-Inferiority — Delta: 15. The significance level for non-inferiority was 0.025; p < 0.001, Hodges-Lehmann estimator; Median Difference (Final Values) = -9, 95% CI 2-sided [-21 to 3]
Statistical Analysis 2: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Superiority; p = 0.175, Hodges-Lehmann estimator — We adjusted for two outcomes for the superiority testing only, using a significance criterion of 0.0125 for each outcome (i.e., 0.025/2, Bonferroni correction), since superiority on either outcome would suffice; Median Difference (Final Values) = -9, 97.5% CI 2-sided [-23 to 5]

3. Secondary Outcome: Time-weighted Pain Score
Description: Postoperative pain was evaluated with numeric rating scores (0-10) at 15-min intervals for the initial two postoperative hours or until discharge, whichever came first. A time-weighted averages pain score is equal to the sum of the portion of each time interval (as a decimal, such as 0.25h) multiplied by the levels of the pain (0-10 numeric rating scores) during the time period divided by 48h.
Time Frame: 15-min interval after surgery until postoperative 2 days or discharge, whichever came first
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
units on a scale | 4.8 (1.8) | 5.2 (1.9)
Statistical Analysis 1: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Non-Inferiority — Delta: 1 The significance level for the non-inferiority test was 0.025; p < 0.001, Regression, Linear — This is a joint hypothesis testing. We tested non-inferiority on both secondary outcomes. If both showed significant non-inferiority, we tested superiority on both outcomes; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.8 to 1]
Statistical Analysis 2: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Superiority; p = 0.094, Regression, Linear — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.4, 97.5% CI 2-sided [-0.8 to 0.1]

4. Secondary Outcome: Opioid-related Side Effects Score POD1 (Postoperative Day 1)
Description: Opioid-Related Symptom Distress Scale (ORSDS) evaluates opioid-related side effects. ORSDS is a 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 12 opioid-related side effects. The mean of the 12 scores are reported with a range from 0-4 where the higher scores mean more opioid-related side effects.
Time Frame: POD1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
score on a scale | 2 [1 to 3] | 2 [1 to 3]

5. Secondary Outcome: Opioid-related Side Effects Score POD2 (Postoperative Day 2)
Description: as for outcome 4
Time Frame: POD2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
score on a scale | 2 [1 to 3] | 2 [1 to 2]

6. Other Pre Specified Outcome: Exploratory Outcome Measurement Patient Satisfaction With Pain Management at Discharge From the Hospital (Numeric Rating System 1-100)
Description: The patient satisfaction with pain management at discharge using (NRS 1-100) or on POD 3 or discharge, whichever comes earlier. The higher score means a better outcome
Time Frame: POD 3 (72 hours) or discharge, whichever comes earlier
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 145 | 142
units on a scale | 78 (22) | 81 (20)

7. Other Pre Specified Outcome: Exploratory Outcome Measurement Quality of Recovery (QoR) Score at 1 Months
Description: Quality of postoperative recovery will be assessed by asking the patient "how have you been feeling during the past 24 hours." Using the Quality of recovery form (QoR15) to document their replies. Quality of recovery (QoR15) score of (0 to 10), where: (0) none of the time (poor) and (10) equal all of the time (excellent). There are a total of 15 questions with each score ranging from 0 to 10. The range of reported total score is 0-150 where higher scores mean better quality of recovery.
Time Frame: At 1 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 137 | 136
units on a scale | 125 (22) | 122 (20)

8. Other Pre Specified Outcome: Exploratory to Measure PDQ (Pain Disability) Using EQ-5D
Description: Using EQ-5D questionnaire for pain disability measurements, at 3 months with the flexibility of +/- 5 days using the EQ-5D questionnaire (0) no pain to (10) worst pain. EQ-5D is a standardized measure of health status developed by EuroQol GROUP
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 127 | 115
units on a scale | 7.0 (2.0) | 7.3 (2.1)

9. Other Pre Specified Outcome: Exploratory to Measure Health-related Quality of Life Using EQ-5D
Description: It is one of several instruments used to verify the quality-adjusted life years associated with a health state. It is defined as a survey instrument for measuring economic preferences for health states based on the assessment of mobility, self-care, usual activities, pain/discomfort and anxiety/depression (5 items in total). Each dimension has 3 levels: 1=no problem, 2=moderate problem, 3=severe problem. The total scores are calculated for each subject.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 143 | 139
units on a scale | 8.6 (2.0) | 9.1 (2.4)

10. Other Pre Specified Outcome: Exploratory Outcome: Chronic Postsurgical Pain at 3 Months (0-10 NRS Scale)
Description: The exploratory outcome chronic postsurgical pain at 3 months was assessed by phone call using a numeric rating scale (0 to 10) where a score of 0 is "no pain" and a score of 10 is "pain as bad as it could be."
Time Frame: at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 122 | 111
units on a scale | 2.6 (.5) | 2.9 (2.9)

11. Other Pre Specified Outcome: Exploratory Outcome: PACU Length of Stay (h)
Description: Postoperative-anesthesia care unit (PACU) length of stay measured how many hours the patient had spent in PACU.
Time Frame: from the time when patients were transferred to the Post-Anesthesia Care Unit to the time when patients were transferred out from the Post-Anesthesia Care Unit.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 149 | 146
hours | 3.6 [2.6 to 5.0] | 3.3 [2.6 to 4.4]

12. Other Pre Specified Outcome: Exploratory Outcome: Number of Patients Who Had Postoperative Nausea and Vomiting in PACU
Description: Postoperative nausea and vomiting was assessed using Postoperative Nursing Progress Record (NPR) - Records nausea vomiting severity as 0=none, 1= mild, 2=moderate, 3= severe.
Time Frame: postoperative time until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 146 | 147
Participants
  None | 91 | 95
  Mild | 27 | 30
  Moderate | 15 | 12
  Severe | 13 | 10

13. Other Pre Specified Outcome: Exploratory Outcome: Postoperative Length of Hospital Stay (Days)
Description: Postoperative length of hospital stay measured how many days the patient had spent in the hospital after surgery.
Time Frame: postoperative time until discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
days | 3 [1 to 5] | 4 [1 to 6]

14. Other Pre Specified Outcome: Exploratory Outcome: Need for Acute Pain Consultation, as Determined by Clinical Need
Description: The outcome measured how many patients needed acute pain consultation after the surgery, as determined by clinical need
Time Frame: postoperative until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 119 | 121
Participants | 16 | 13

15. Post Hoc Outcome: Exploratory Outcome: Number of Participants With Postoperative Acetaminophen Use
Description: This outcome measured how many patients used acetaminophen during the 48 hours after the surgery
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 141 | 136

16. Post Hoc Outcome: Exploratory Outcome: the Number of Patients Who Had Postoperative Gabapentin
Description: This outcome measured how many patients used postoperative gabapentin during the 48 hours after the surgery.
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 59 | 59

17. Post Hoc Outcome: Exploratory Outcome: the Number of Patients Who Had Postoperative Tramadol
Description: This outcome measured how many patients used postoperative tramadol during the 48 hours after the surgery.
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 1 | 7

18. Post Hoc Outcome: Exploratory Outcome: the Number of Patients Who Had Postoperative Ketorolac Within 48 Hours
Description: This outcome measured how many patients used postoperative ketorolac during the 48 hours after the surgery.
Time Frame: within 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 38 | 38

19. Post Hoc Outcome: Exploratory Outcome: the Number of Patients Who Had Postoperative Suboxone Within 48 Hours
Description: This outcome measured how many patients used postoperative suboxone during the 48 hours after the surgery.
Time Frame: within 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 0 | 0

20. Post Hoc Outcome: Exploratory Outcome: the Number of Patients Who Had Postoperative PCA (Patient-controlled Analgesia) Use Within 48h
Description: This outcome measured how many patients used postoperative patient-controlled analgesia during the 48 hours after the surgery.
Time Frame: within 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
Participants | 90 | 81

21. Post Hoc Outcome: Secondary Outcome: 24-h Opioid Consumption
Description: This outcome measured how many postoperative opioids (mg in morphine equivalents) patients used during the 24 hours after the surgery.
Time Frame: within 24 hours after the surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
mg | 47 [26 to 68] | 45 [33 to 81]
Statistical Analysis 1: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Non-Inferiority — Delta: 9; significance level was 0.025; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 2: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Superiority; p = 0.171, Wilcoxon sum rank test — [p-value comment as in outcome 2, analysis 2]; Median Difference (Final Values) = -0.1, 97.5% CI 2-sided [-0.3 to 0.1]

22. Post Hoc Outcome: Secondary Outcome: 24h Time-weighted Average Pain Score
Description: Pain score is a 10 point scale score where the higher means more pain.
Time Frame: within 24 hours after the surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
Number analyzed (Participants) | 150 | 149
score on a scale | 4.8 (1.9) | 5.3 (2.0)
Statistical Analysis 1: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Non-Inferiority — Delta: 1 significance level: 0.025; p < 0.001, Regression, Linear; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to -0.1]; The superiority test (this is a joint-hypothesis testing) showed a mean difference of -0.5 between treatment and control group with 97.5% CI of (-1.0, 0.0) and p-value of 0.025. The significance level was 0.025
Statistical Analysis 2: Comparison: Spine Surgery Analgesic Pathway vs Usual Care; Test type: Superiority; p = 0.025, Regression, Linear — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.5, 97.5% CI 2-sided [-1.0 to 0.0]

ADVERSE EVENTS:
Time Frame: within 3 months since the onset of treatment
Arm/Group | Spine Surgery Analgesic Pathway | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/149
Other Adverse Events (participants affected / at risk) | 0/150 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02887404/Prot_SAP_000.pdf